CLINICAL TRIAL: NCT06123299
Title: A Randomised, Partly-blinded Investigation to Evaluate the Clinical Performance and Safety of pHyph in Adult Women With Bacterial Vaginosis Compared With an Untreated Control Group
Acronym: Nefertiti 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gedea Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL3-2
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pHyph treatment (Active Comparator): Initial treatment with pHyph vaginal tablet once daily during 6 consecutive days
  Interventions: Device: pHyph
- No treatment (No Intervention): No initial treament during the first 7 days of the study

INTERVENTIONS:
Device: pHyph — vaginal tablet
  Arms: pHyph treatment

SUMMARY:
This is a randomised, parallel group, partly blinded investigation to evaluate the clinical performance and safety of pHyph in adult women with bacterial vaginosis. Patients will be randomised to active treatment or no treatment (untreated controls) in a 1:1 ratio. The Investigators carrying out the gynaecological assessments will be blinded. Patients will not be blinded.

The population of this investigation will consist of post-menarchal, pre-menopausal females 18 years or older seeking treatment for BV symptoms ("fishy smell", irritation and burning).

Approximately 82-92 patients will be recruited and randomised. BV will be diagnosed according to Amsel's criteria, defined as having at least 3 of the 4 criteria.

Active treatment (from the start of the investigation) will be compared to no treatment at day 7 after screening (primary endpoint). Clinical cure rate on Day 7 is defined as the absence of all of the following 3 Amsel criteria:

* Thin, white, yellow, homogeneous discharge.
* Clue cells on microscopy (>20% of epithelial cells).
* Release of a "fishy odour", i.e., a positive "whiff test" when alkali (10% KOH solution) is added.

Patients receiving rescue treatment before Day 7 will be considered as treatment failures.

Patients in the "no treatment group" will receive pHyph as rescue treatment if they are not cured day 7. They will thereafter follow the same scheme as the patients starting with pHyph treatment.

After the initial pHyph treatment, daily during 6 days, patients will continue with pHyph twice weekly until day 25 when an additional assessment will be performed. If the patients are cured, they will continue to receive pHyph as preventive treatment during 6 weeks and possible BV recurrences will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the clinical investigation, and to comply with all clinical investigation requirements.
2. Adult, post-menarchal, pre-menopausal women aged 18 years or older.
3. Diagnosis of BV according to Amsel's criteria, defined as having at least 3 of the 4 following criteria:

   * Thin, white, yellow, homogeneous discharge.
   * Clue cells on microscopy (>20% of epithelial cells).
   * pH of vaginal fluid >4.5.
   * Release of "fishy odour", i.e., a positive "whiff test" when alkali (10% KOH solution) is added. This symptom must be present.
4. Negative urine pregnancy test at screening.
5. Willing to refrain from using any intravaginal products (e.g., contraceptive creams, gels, foams, sponges, lubricants or tampons, etc.) until Day 7 and the following 24 hours after each pHyph administration during weekly treatment.
6. Willing to use condoms during any sexual intercourse with a male sexual partner until the initial pHyph treatment is completes. For patients starting with pHyph on Day 0, this means from Visit 1 (Day 0) until Visit 2 (Day 7). For patients that do not receive any treatment between Day 0 and Day 7, this means from Visit 1 (Day 0), and if they receive pHyph from Day 7, until their Visit 2 (Day 14).
7. Willing to use a method of contraception, e.g., condoms, hormonal contraception (oral, injectable, implantable, intravaginal, or transdermal), intrauterine device (IUD) or intrauterine hormone-releasing system (IUS), during any sexual intercourse that might result in pregnancy from Visit 2 (Day 7 or 14) until Visit 4 (70-77 days) to prevent pregnancy.

Exclusion Criteria:

1. Patients with known or apparent signs of other infectious causes of vaginitis (e.g., vulvovaginal candidiasis, Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis, Herpes simplex, or human papillomavirus) at screening.
2. History of or presence at screening (Day 0) of any other clinically significant disease or disorder, medical/surgical procedure, or trauma, which, in the opinion of the Investigator, may either put the patient at risk because of participation in the clinical investigation, or influence the results or the patient's ability to participate in the clinical investigation.
3. Anticipated menstruation during the initial daily treatment period (Day 0 until Day 5).
4. Patients who are pregnant or breastfeeding.
5. Patients who are planning to conceive within the 70-77 days of the investigation.
6. Patients who were treated for BV within the 14 days preceding screening.
7. Patients who are currently receiving antibiotic therapy unrelated to BV or have received antibiotic therapy within the 14 days preceding screening.
8. Patients who have used any pH-modifying vaginal products within the 14 days preceding screening.
9. Patients who have received an investigational drug in a clinical trial within 30 days prior to screening.
10. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, to any of the product components.
11. The Investigator considers the patient unlikely to comply with clinical investigation procedures, restrictions and requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate on Day 7 | 7 days
  Defined as the absence of all of the following 3 Amsel criteria:
  * Thin, white, yellow, homogeneous discharge.
  * Clue cells on microscopy (>20% of epithelial cells).
  * Release of a "fishy odour", i.e., a positive "whiff test" when alkali (10% potassium hydroxide [KOH] solution) is added.

SECONDARY OUTCOMES:
Proportion of patients that do not have the symptom "fishy odour" on Days 1 to 7 after start of treatment, compared to Day 0, measured by using a patient questionnaire administered via mobile application. | 7 days
Proportion of patients that do not have the symptom "fishy odour" on Day 7 after start of treatment, compared to Day 0, as assessed by the Investigator as part of the Amsel criteria. | 7 days
Proportion of patients having a reduction in each of 3 BV symptoms scores on Days 1 to 7 after start of treatment, compared to Day 0, measured by using a patient questionnaire administered via mobile application. | 7 days
Safety and local tolerability of pHyph for patients receiving daily treatment for 6 days, based on the reported treatment-emergent AEs up until Day 7 after start of treatment. | 7 days
Clinical cure rate on Day 7 after start of treatment, defined as clinical cure according to secondary endpoint 1 and Nugent score <4, i.e., both criteria have to be fulfilled. | 7 days
Clinical cure rate on Day 7 after start of treatment, defined as Nugent score <4. | 7 days
Usability measured using a patient questionnaire administered via mobile application on Day 7 and Day 25. | Day 7 and 25
Difference between Day 0, Day 7, and Day 25 after start of treatment in the occurrence of anaerobic vaginal dysbiosis, as assessed by analysis of the vaginal microbiome. | Day 25
Difference between Day 0, Day 7, and Day 25 after start of treatment in the occurrence of vaginal yeasts, as assessed by analysis of the vaginal microbiome. | Day 25
For the subgroup of patients with a Nugent score ≥7 on Day 0: Primary endpoint and secondary endpoints 1-4, and 6. | 7 days
Proportion of patients that do not have the symptom "fishy odour" on Day 25 after start of treatment, as assessed by the Investigator as part of the Amsel criteria. | 25 days
Proportion of patients that do not have the symptom fishy "odour" on Day 25 after start of treatment, as assessed by the Investigator as part of the Amsel criteria, and Nugent score <4, i.e., both criteria have to be fulfilled. | 25 days
Clinical cure rate on Day 25 after start of treatment, defined as clinical cure according to the primary endpoint. | 25 days
Clinical cure rate on Day 25 after start of treatment, defined as clinical cure according to the primary endpoint and Nugent score <4, i.e., both criteria have to be fulfilled. | 25 days
Proportion of patients having a reduction in pH on Day 7 after start of treatment compared to Day 0. | 7 days
Recurrence from day 25, as defined by vaginal dysbiosis | 70 days
  Difference between Visit 3, Day 55, and Visit 4, or day of possible recurrence confirmation, respectively, in the occurrence of anaerobic vaginal dysbiosis as assessed by analysis of the vaginal microbiome, in patients starting with active treatment on Day 0 and patients starting with active treatment on Day 7, respectively and together.
Recurrence from day 7, as defined by clinical assessment | 70 days
  Recurrence rate from Day 7 in patients starting with active treatment on Day 0 (active treatment group) and patients starting with active treatment on Day 7 (no initial treatment group), respectively and together.
  1. Defined as the proportion of patients diagnosed with BV according to Amsel's criteria, defined as having at least 3 of the 4 criteria.
  2. Defined as the proportion of patients diagnosed with BV according to Amsel's criteria, defined as having at least 3 of the 4 criteria, and according to Nugent score defined as having a score of ≥7, i.e., both criteria have to be fulfilled.
  3. Defined as the presence of "fishy odour" reported by the patient in connection with reporting of the confirmed recurrence as defined in secondary endpoints 17a and 17b.
Recurrence from day 25, as defined by clinical assessment | 70 days
  Recurrence rate from Day 25 in patients starting with active treatment on Day 0 (active treatment group) and patients starting with active treatment on Day 7 (no initial treatment group), respectively and together.
  1. Defined as the proportion of patients diagnosed with BV according to Amsel's criteria, defined as having at least 3 of the 4 criteria.
  2. Defined as the proportion of patients diagnosed with BV according to Amsel's criteria, defined as having at least 3 of the 4 criteria, and according to Nugent score defined as having a score of ≥7, i.e., both criteria have to be fulfilled.
  3. Defined as the presence of "fishy odour" reported by the patient in connection with reporting of the confirmed recurrence as defined in secondary endpoints 18a and 18b.
Safety and local tolerability for patients receiving preventive treatment: | 70 days
  a. Based on reported treatment-emergent adverse events (AEs) from Visit 3 up until Visit 4.
Safety and local tolerability for patients receiving preventive treatment: | 70 days
  b. Based on signs of erythema, oedema and excoriation on the vaginal mucosa, according to a scoring scale (0-3), assessed at Visit 1, 2, 3, and 4/or day of possible recurrence confirmation.

OTHER OUTCOMES:
Exploratory endpoints 1 | 70 days
  The results from the analysis of the vaginal microbiome on Days 0, 7, 25, and 70 (active treatment group) or Days 7, 14, 32 and 77 (no initial treatment group), and/or day of BV recurrence confirmation, performed by a central laboratory, will be evaluated further on an exploratory basis.
Exploratory endpoints 2 | 70 days
  The results from the analysis of the vaginal microbiome on Day 7 after the start of rescue treatment will also be evaluated on an exploratory basis. For this patient group, the frequency of self-reported BV recurrence will also be evaluated.
Exploratory endpoints 3 | 70 days
  For patients receiving rescue treatment, treatment usability will be measured using the same questionnaire as specified in secondary endpoint 7

CONTACTS AND LOCATIONS:
Overall Officials: Aino Fianu Jonasson, Ass. Prof., Principal Investigator — Karolinska Institute, Stockholm
Locations (5):
- Sweden (5):
  - CTC, Ebbe Park, Linköping
  - CTC GoCo, Mölndal
  - CTC, Karolinska, Solna
  - Kvinnoforskningsenheten, KS Huddinge, Stockholm
  - CTC MTC, Uppsala

IPD SHARING:
Plan to Share IPD: No